CLINICAL TRIAL: NCT06075134
Title: EMG-guided Botox Injection Versus Conventional Injection in Yonsei Point in Gummy Smile Patients: A Randomized Clinical Trial
Brief Title: EMG-guided Botox Injection Versus Conventional Botox Injection in Gummy Smile Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherry Fayez Akhnokh, Periodontology Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFAkhnokh
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Excessive Gingival Display
MeSH Terms: interventions — Botulinum Toxins, Type A; Botulinum Toxins; Electromyography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG-guided Botox injection (Experimental): Botox injection in patients with gummy smile will be done under electromyography guidance to target the most hyperactive and effective muscle that is the chief factor causing the condition.
  Interventions: Procedure: Botox injection; Device: EMG; Drug: Zinc Supplement
- Conventional Botox injection in Yonsei point (Active Comparator): Conventional injection of Botox is located in Yonsei point, which is the center of a triangle formed by the convergence of Levator labii superioris alaeque nasi (LLSAN), levator labii superioris (LLS), zygomaticus minor (ZMn), muscles, and is located 1 cm lateral to the ala of the nose horizontally and 3 cm above the lip line vertically.
  Interventions: Procedure: Botox injection; Drug: Zinc Supplement

INTERVENTIONS:
Procedure: Botox injection — Botox injection
  Other Names: Botulinum toxin injection
Device: EMG — Quantitative Electromyography
  Other Names: Electromyography
  Arms: EMG-guided Botox injection
Drug: Zinc Supplement — To increase efficacy of Botox
  Other Names: Zinc supplement in the form of tablets

SUMMARY:
The goal of this clinical trial is to compare the effect of EMG-guided Botox injection with conventional Botox injection in Yonsei point, in patients with excessive gingival display.

The main question it aims to answer is:

• Does the use of electromyography (EMG) as a guide during Botox injection for patients with gummy smile has better effect than conventional injection in Yonsei point?

Participants will be randomized in equal proportions between intervention and control groups.

* Preoperative assessment of amount of gingival display, lip length (philtrum and vermilion length), and smile type.
* For the intervention group, EMG readings will be done in Clinical Neurophysiology Department, Kasr Al-Ainy Hospital EMG-guided Botox injection (Intervention group). Conventional Botox injection in Yonsei point (Control group).

ELIGIBILITY:
Inclusion Criteria:

* Patients with excessive gingival display.
* Patients with esthetic concerns.
* Patients with mild to moderate VME (vertical maxillary excess).
* Normal clinical crown dimensions.
* Patients aged 18 to 50.
* Systemically healthy patients.
* Non-smokers.

Exclusion Criteria:

* Patients with severe VME (vertical maxillary excess).
* Pregnant and breastfeeding women.
* Patients with gingival inflammation and/or enlargement.
* Inflammation or infection at the site of injection.
* Patients with known allergy to any of the components of Botox (i.e., saline, human albumin, lactose and sodium succinate).
* Patients using anticholinesterase or other agents affecting neuromuscular transmission.
* Psychologically unstable patients or those who have unrealistic expectations and questionable motives.
* Patients with neuromuscular disorders (e.g., myasthenia gravis, Eaton-Lambert syndrome).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in amount of gingival display | Baseline, One-week, One-month, three-months, and six-months follow-up
  Will be measured using ruler in mm.

SECONDARY OUTCOMES:
Quantitative EMG | Baseline, One-week and six-months follow-up
  Will be measured using EMG in mv.
Patient satisfaction | Baseline, One-week, One-month, three-months, and six-months follow-up
  Will be assessed using questionnaire, on a scale from 1 to 5, where 1 is completely not satisfied and 5 is completely satisfied.
Post-operative pain | Baseline, One-week, and One-month follow-up
  Will be measured using visual analogue scale (VAS) from 1 to 10.
Smile type | Baseline, One-week, One-month, three-months, and six-months follow-up
  Qualitative, by Rubin (1974). Smile is classified into 1. Corner of the mouth (Mona Lisa) smile, 2. Canine Smile, and 3. Full denture smile
Change in lip length | Baseline, One-week, One-month, three-months, and six-months follow-up
  Will be measured using UNC (University of North Carolina) -15 periodontal probe in mm.
Esthetics (Symmetry) for operators | Baseline, One-week, One-month, three-months, and six-months follow-up
  Will be measured using 5-point Likert scale, where 1 is significantly asymmetrical and 5 is completely symmetrical.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Fayez Akhnokh, BSc, Principal Investigator — Cairo University; Noha Ghallab, PhD, Study Director — Cairo University; Nesma Shemais, PhD, Study Chair — Cairo University